CLINICAL TRIAL: NCT06842095
Title: Investigating the Effects of Beta Transcranial Stimulation to Advance Stroke Rehabilitation
Brief Title: Investigating the Effects of Transcranial Stimulation to Advance Stroke Rehabilitation
Acronym: T-STAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PID17878
Record Dates: First submitted 2024-10-23; First posted 2025-02-24 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-07

CONDITIONS: Stroke; Upper Limb Function
Keywords: Non-Invasive Brain Stimulation; Stroke; Upper Limb; Electroencephalography; Transcranial Alternating Current Stimulation; Beta Oscillations
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: There will be two experimenters: one delivering the stimulation, who will NOT be blinded and one who will be taking behavioural measures and communicating with the participant who WILL be blinded to stimulation condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Stimulation (beta-tACS) (Experimental): Participants will receive one session of active stimulation (beta-tACS) to the ipsilesional hemisphere. The electrode montage will include one electrode positioned on the scalp over the left or right motor cortex (either C3 or C4 using the international 10-20 EEG system), depending on the location of the stroke, and a second electrode over posterior area (Pz). A low intensity of stimulation (max. 4 mA peak to peak amplitude) will be used for up to 30 minutes in total (delivered in short bouts of up to 5 seconds based on the timing of movement of the upper limb).
  Interventions: Other: Transcranial Alternating Current Stimulation (beta-tACS)
- Sham Stimulation (tACS) (Sham Comparator): Participants will receive one session of sham stimulation. The electrode placement will be the same as for the experimental condition, but duration or timing of stimulation will be insufficient to induce intended brain rhythm changes.
  Interventions: Other: Transcranial Alternating Current Stimulation (sham)

INTERVENTIONS:
Other: Transcranial Alternating Current Stimulation (beta-tACS) — The study intervention is transcranial alternating current stimulation (tACS).
  The electrode montage will include one electrode positioned on the scalp over the left or right motor cortex (either C3 or C4 using the international 10-20 EEG system), depending on the location of the stroke, and a second electrode over posterior area (Pz). A low intensity of stimulation (max. 4 mA peak to peak amplitude) will be used for up to 30 minutes in total (delivered in short bouts of up to 5 seconds based on the timing of movement of the upper limb).
  Other Names: Non Invasive Brain Stimulation; beta tACS
  Arms: Active Stimulation (beta-tACS)
Other: Transcranial Alternating Current Stimulation (sham) — The comparator is sham stimulation. Stimulation is delivered for a very short duration or timed in such a way relative to movement to mimic the scalp sensations of the active stimulation without delivering stimulation that would be anticipated to impact relevant brain activity rhythms.
  Other Names: tACS (sham)
  Arms: Sham Stimulation (tACS)

SUMMARY:
Non-invasive brain stimulation (NIBS) has the potential to boost rehabilitation after stroke by creating a 'pro-plastic' environment, where the brain is more adaptable in response to movement (motor) training. However, responses to classical NIBS protocols are highly variable.

Movement-related changes in specific brain rhythms have previously been shown to be related to recovery of hand/arm function after a stroke. The investigators propose to use NIBS to target movement-related activity in the beta band (13-30Hz) within the motor cortical regions of the brain. The investigators will use a type of NIBS called transcranial alternating current stimulation (tACS), which uses a sinusoidally-varying electrical current where the stimulation frequency is determined to be relevant to the underlying brain rhythms of interest, and the stimulation timed to coincide with specific phases of the hand/arm movement.

The primary aim is to investigate whether beta-tACS improves upper limb movement in stroke survivors.

DETAILED DESCRIPTION:
Stroke is a leading cause of death and long-term disability worldwide. More than 70% of stroke survivors experience motor impairments, often resulting in difficulties in daily activities, such as walking, reaching and grasping objects. Regaining upper-limb motor function is key to quality of life and for reducing the high annual costs due to stroke.

Research indicates that upper-limb motor function recovery depends on the plasticity of neural circuits controlling movement. Beta activity (β, ~13-30 Hz) in the sensorimotor cortex has been associated with brain plasticity and has been proposed to play a pivotal role in human movement and movement disorders. This activity attenuates during movement execution, known as event-related desynchronization (β-ERD), and temporarily increases after the end of movement, known as event-related synchronization (β-ERS).

β-ERD and β-ERS are reliably observed during active and passive movement, movement imagination and movement observation. Changes in movement-related β-ERD and β-ERS have been linked to motor learning, and motor dysfunction in neurological conditions, such as stroke. Studies have shown that stroke survivors with upper limb impairments exhibit significantly lower beta activity compared to healthy individuals, and recovery-related improvements in motor function are accompanied by increases in both sensorimotor β-ERD and β-ERS.

Therefore, modulation of movement-related beta activity (i.e., β-ERD and β-ERS) holds great promise for promoting motor function after stroke. Non-invasive brain stimulation (NIBS) can be applied during movements to increase plasticity and enhance motor learning and function. However, prior studies have delivered NIBS using a relatively broad approach; modulating general cortical excitability rather than enhancing specific endogenous oscillations in the brain. Transcranial alternating current stimulation (tACS) is a safe and well-tolerated type of NIBS which provides an option for modulating specific frequencies of brain oscillations by delivering a low-intensity sinusoidal electrical current to the brain at a specific frequency.

Therefore, this study will deliver beta-tACS to the ipsilesional motor cortex (M1) aiming to modulate sensorimotor beta activity during upper limb movement in stroke survivors. This study will investigate whether functionally timed beta-tACS has the potential to enhance motor recovery, by assessing whether stimulation delivered at the end of the movement improves upper limb movement (accuracy, smoothness and hand function) and increases the modulation of beta activity. Additionally, the investigators will evaluate whether the effectiveness of the stimulation relates to baseline neuroimaging and neurophysiological measures. Identifying correlates of intervention responsiveness will help future studies to target patients who are most likely to benefit.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Aged 18 years or above.
* Clinical diagnosis of stroke affecting the upper limb, with sufficient ability to perform the upper limb reaching task.
* At least 3 months post-stroke and discharged from inpatient care.

Exclusion Criteria:

* Inability to follow task instructions.
* Other neurological condition affecting movement (e.g. Parkinson's Disease, Multiple Sclerosis).
* Standard contraindications to non-invasive brain stimulation (TMS, tACS). including (but not limited to) the presence of intracranial metallic or magnetic hardware, seizures, pregnancy, and the presence of a pacemaker or other stimulators/implants.
* Insufficient verbal and written English to comprehend the study and provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Reaching Performance | From the first stimulation session to the completion of the third and final session, an average of 1 month
  Performance on the reaching task, assessed using a motion sensor as the error (deviation from the ideal path) in cubic centimeters. Higher numbers indicate worse error/reaching performance.

SECONDARY OUTCOMES:
Movement-related Brain Rhythms | From the first stimulation session to the completion of the third and final session, an average of 1 month
  Movement-related beta activity measured using electroencephalography (EEG), as power in decibels. Higher values indicate stronger (better) movement-related beta activity.
Hand Function | From the first stimulation session to the completion of the third and final session, an average of 1 month
  Change in hand function measured with the Box and Blocks Test from pre-stimulation to post-stimulation. Box and blocks test performance is measured as the number of blocks moved with the affected hand in 1 minute, higher numbers indicate better hand function.

OTHER OUTCOMES:
Smoothness of reaching movement (peaks) | From the first stimulation session to the completion of the third and final session, an average of 1 month
  Smoothness of reaching movement assessed using a motion sensor as the number of peaks (number). Higher values indicate worse smoothness of reaching movement.
Smoothness of reaching movement (arrest periods) | From the first stimulation session to the completion of the third and final session, an average of 1 month
  Smoothness of reaching movement assessed using a motion sensor as the time of arrest periods (seconds). Higher numbers indicate worse smoothness of movement.
Smoothness of reaching movement (Jerk) | From the first stimulation session to the completion of the third and final session, an average of 1 month
  Smoothness of reaching movement assessed using a motion sensor as the jerk metric (time rate of change in acceleration) in centimeters per second. Lower values indicate better smoothness of reaching movement.
Brain Structure at baseline (grey matter volume) | baseline
  Brain structure measured with magnetic resonance imaging at baseline as the volume of grey matter in the motor-related areas of the ipsilesional hemisphere of the brain. Higher numbers indicate greater grey matter (brain) volume.
Brain Function at Baseline (connectivity) | baseline
  Brain function measured with resting state functional magnetic resonance imaging at baseline. Higher numbers indicate greater functional brain connectivity.
Brain Function (neurochemicals) at Baseline | baseline
  Brain function measured with magnetic resonance spectroscopic imaging as the concentration of neurochemicals GABA and Glutamate in the sensorimotor regions of interest. Higher numbers indicate a greater neurochemical concentration.
Corticospinal tract integrity at Baseline | baseline
  Corticospinal tract integrity measured as the presence or absence of a motor evoked potential in the affected upper limb using transcranial magnetic stimulation at baseline (binary yes=1, no-0). A score of 1(yes) indicates a (at least partially) intact corticospinal tract.
Motor Ability at Baseline (Action Research Arm Test) | baseline
  Motor ability assessed with the Action Research Arm Test, score 0-57. Higher numbers indicate better upper limb motor ability
Motor Impairment at Baseline (Fugl Meyer Assessment) | baseline
  Upper Limb Motor impairment assessed with the Fugl Meyer Assessment, score 0-66. Higher numbers indicate less upper limb motor impairment
Brain Structure at baseline (grey matter damage) | baseline
  Brain structure measured with magnetic resonance imaging at baseline as the percentage (%) of regions (parcels) damaged by the lesion. Higher numbers indicate greater grey matter (brain) damage.
Brain Structure at baseline (white matter damage) | baseline
  Brain structure measured with magnetic resonance imaging at baseline as the percentage (%) of regions (tracts) disconnected due to the lesion. Higher numbers indicate greater white matter (brain) damage.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte J Stagg, PhD, Principal Investigator — University of Oxford; Catharina Zich, PhD, Study Director — University of Oxford
Locations (1):
- Oxford Centre for Functional MRI of the Brain (FMRIB), Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on reasonable request to the Chief Investigator, Dr Fleming or Dr Zich.
Supporting Information: Analytic Code
Time Frame: After publication of the results. There is no definitive end date

REFERENCES:
- [Background] Wischnewski M, Schutter DJLG, Nitsche MA. Effects of beta-tACS on corticospinal excitability: A meta-analysis. Brain Stimul. 2019 Nov-Dec;12(6):1381-1389. doi: 10.1016/j.brs.2019.07.023. Epub 2019 Jul 28. PMID 31405789
- [Background] Toledo DR, Manzano GM, Barela JA, Kohn AF. Cortical correlates of response time slowing in older adults: ERP and ERD/ERS analyses during passive ankle movement. Clin Neurophysiol. 2016 Jan;127(1):655-663. doi: 10.1016/j.clinph.2015.05.003. Epub 2015 May 9. PMID 26024982
- [Background] Tang CW, Hsiao FJ, Lee PL, Tsai YA, Hsu YF, Chen WT, Lin YY, Stagg CJ, Lee IH. beta-Oscillations Reflect Recovery of the Paretic Upper Limb in Subacute Stroke. Neurorehabil Neural Repair. 2020 May;34(5):450-462. doi: 10.1177/1545968320913502. Epub 2020 Apr 23. PMID 32321366
- [Background] Stancak A Jr, Pfurtscheller G. Desynchronization and recovery of beta rhythms during brisk and slow self-paced finger movements in man. Neurosci Lett. 1995 Aug 18;196(1-2):21-4. doi: 10.1016/0304-3940(95)11827-j. PMID 7501247
- [Background] Stagg CJ, Bachtiar V, Johansen-Berg H. The role of GABA in human motor learning. Curr Biol. 2011 Mar 22;21(6):480-4. doi: 10.1016/j.cub.2011.01.069. Epub 2011 Mar 3. PMID 21376596
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Pogosyan A, Gaynor LD, Eusebio A, Brown P. Boosting cortical activity at Beta-band frequencies slows movement in humans. Curr Biol. 2009 Oct 13;19(19):1637-41. doi: 10.1016/j.cub.2009.07.074. Epub 2009 Oct 1. PMID 19800236
- [Background] Pfurtscheller G, Neuper C, Brunner C, da Silva FL. Beta rebound after different types of motor imagery in man. Neurosci Lett. 2005 Apr 22;378(3):156-9. doi: 10.1016/j.neulet.2004.12.034. Epub 2005 Jan 8. PMID 15781150
- [Background] Pfurtscheller G, Berghold A. Patterns of cortical activation during planning of voluntary movement. Electroencephalogr Clin Neurophysiol. 1989 Mar;72(3):250-8. doi: 10.1016/0013-4694(89)90250-2. PMID 2465128
- [Background] Peter J, Ferraioli F, Mathew D, George S, Chan C, Alalade T, Salcedo SA, Saed S, Tatti E, Quartarone A, Ghilardi MF. Movement-related beta ERD and ERS abnormalities in neuropsychiatric disorders. Front Neurosci. 2022 Nov 23;16:1045715. doi: 10.3389/fnins.2022.1045715. eCollection 2022. PMID 36507340
- [Background] Owolabi MO, Thrift AG, Mahal A, Ishida M, Martins S, Johnson WD, Pandian J, Abd-Allah F, Yaria J, Phan HT, Roth G, Gall SL, Beare R, Phan TG, Mikulik R, Akinyemi RO, Norrving B, Brainin M, Feigin VL; Stroke Experts Collaboration Group. Primary stroke prevention worldwide: translating evidence into action. Lancet Public Health. 2022 Jan;7(1):e74-e85. doi: 10.1016/S2468-2667(21)00230-9. Epub 2021 Oct 29. PMID 34756176
- [Background] Neuper C, Wortz M, Pfurtscheller G. ERD/ERS patterns reflecting sensorimotor activation and deactivation. Prog Brain Res. 2006;159:211-22. doi: 10.1016/S0079-6123(06)59014-4. PMID 17071233
- [Background] Muller-Putz GR, Zimmermann D, Graimann B, Nestinger K, Korisek G, Pfurtscheller G. Event-related beta EEG-changes during passive and attempted foot movements in paraplegic patients. Brain Res. 2007 Mar 16;1137(1):84-91. doi: 10.1016/j.brainres.2006.12.052. Epub 2006 Dec 22. PMID 17229403
- [Background] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Background] Lyle RC. A performance test for assessment of upper limb function in physical rehabilitation treatment and research. Int J Rehabil Res. 1981;4(4):483-92. doi: 10.1097/00004356-198112000-00001. No abstract available. PMID 7333761
- [Background] Liepert J, Miltner WH, Bauder H, Sommer M, Dettmers C, Taub E, Weiller C. Motor cortex plasticity during constraint-induced movement therapy in stroke patients. Neurosci Lett. 1998 Jun 26;250(1):5-8. doi: 10.1016/s0304-3940(98)00386-3. PMID 9696052
- [Background] Liepert J, Bauder H, Wolfgang HR, Miltner WH, Taub E, Weiller C. Treatment-induced cortical reorganization after stroke in humans. Stroke. 2000 Jun;31(6):1210-6. doi: 10.1161/01.str.31.6.1210. PMID 10835434
- [Background] Lawrence ES, Coshall C, Dundas R, Stewart J, Rudd AG, Howard R, Wolfe CD. Estimates of the prevalence of acute stroke impairments and disability in a multiethnic population. Stroke. 2001 Jun;32(6):1279-84. doi: 10.1161/01.str.32.6.1279. PMID 11387487
- [Background] Kulasingham JP, Brodbeck C, Khan S, Marsh EB, Simon JZ. Bilaterally Reduced Rolandic Beta Band Activity in Minor Stroke Patients. Front Neurol. 2022 Mar 28;13:819603. doi: 10.3389/fneur.2022.819603. eCollection 2022. PMID 35418932
- [Background] Koganemaru S, Mima T, Thabit MN, Ikkaku T, Shimada K, Kanematsu M, Takahashi K, Fawi G, Takahashi R, Fukuyama H, Domen K. Recovery of upper-limb function due to enhanced use-dependent plasticity in chronic stroke patients. Brain. 2010 Nov;133(11):3373-84. doi: 10.1093/brain/awq193. Epub 2010 Aug 5. PMID 20688810
- [Background] Kilavik BE, Zaepffel M, Brovelli A, MacKay WA, Riehle A. The ups and downs of beta oscillations in sensorimotor cortex. Exp Neurol. 2013 Jul;245:15-26. doi: 10.1016/j.expneurol.2012.09.014. Epub 2012 Sep 27. PMID 23022918
- [Background] Joundi RA, Jenkinson N, Brittain JS, Aziz TZ, Brown P. Driving oscillatory activity in the human cortex enhances motor performance. Curr Biol. 2012 Mar 6;22(5):403-7. doi: 10.1016/j.cub.2012.01.024. Epub 2012 Feb 2. PMID 22305755
- [Background] Herrmann CS, Rach S, Neuling T, Struber D. Transcranial alternating current stimulation: a review of the underlying mechanisms and modulation of cognitive processes. Front Hum Neurosci. 2013 Jun 14;7:279. doi: 10.3389/fnhum.2013.00279. eCollection 2013. PMID 23785325
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Duncan PW, Bode RK, Min Lai S, Perera S; Glycine Antagonist in Neuroprotection Americans Investigators. Rasch analysis of a new stroke-specific outcome scale: the Stroke Impact Scale. Arch Phys Med Rehabil. 2003 Jul;84(7):950-63. doi: 10.1016/s0003-9993(03)00035-2. PMID 12881816
- [Background] Demeyere N, Riddoch MJ, Slavkova ED, Bickerton WL, Humphreys GW. The Oxford Cognitive Screen (OCS): validation of a stroke-specific short cognitive screening tool. Psychol Assess. 2015 Sep;27(3):883-94. doi: 10.1037/pas0000082. Epub 2015 Mar 2. PMID 25730165
- [Background] Chalard A, Amarantini D, Tisseyre J, Marque P, Gasq D. Spastic co-contraction is directly associated with altered cortical beta oscillations after stroke. Clin Neurophysiol. 2020 Jun;131(6):1345-1353. doi: 10.1016/j.clinph.2020.02.023. Epub 2020 Mar 19. PMID 32304849
- [Background] Bachtiar V, Near J, Johansen-Berg H, Stagg CJ. Modulation of GABA and resting state functional connectivity by transcranial direct current stimulation. Elife. 2015 Sep 18;4:e08789. doi: 10.7554/eLife.08789. PMID 26381352
- [Background] Bachtiar V, Johnstone A, Berrington A, Lemke C, Johansen-Berg H, Emir U, Stagg CJ. Modulating Regional Motor Cortical Excitability with Noninvasive Brain Stimulation Results in Neurochemical Changes in Bilateral Motor Cortices. J Neurosci. 2018 Aug 15;38(33):7327-7336. doi: 10.1523/JNEUROSCI.2853-17.2018. Epub 2018 Jul 20. PMID 30030397